CLINICAL TRIAL: NCT03960736
Title: COMPARISON OF CONTINUOUS ERECTOR SPINAE PLANE BLOCK AND THORACIC EPIDURAL ANALGESIA FOR POSTOPERATİVE ANALGESIA MANAGEMENT FOLLOWING VIDEO ASSISTED THORACIC SURGERY
Brief Title: Continuous Erector Spinae Plane Block or Thoracic Epidural Analgesia Following Video Assisted Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Mega Hospital Complex
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Lung Diseases
Keywords: Video assisted thoracic surgery; Postoperative pain management; Erector spina plane block; Thoracic epidural analgesia
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: Sixty patients aged 18-65 years old with American Society of Anesthesiologists (ASA) classification I-II and scheduled for VATS under general anesthesia will be included in the study. Patients with a history of bleeding diathesis, receiving anticoagulant treatment, known local anesthetics and opioid allergy, infection of the skin at the site of the needle puncture, pregnancy or lactation, and patients who do not accept the procedure will be excluded from the study. Randomization will be achieved using a randomizing computer program. Patients will be randomly divided into two groups (Group A = ESP group, Group B = TEA group) including 25 patients each, before entering the operating room.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes Assessor and the patient will be blinded to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ESPB = Erector spinae plane block group (Active Comparator): ESP block (Group ESP) will be performed in the preoperative block room.A continuous infusion of 0.125% bupivacaine at the rate of 4 ml/h infusion dose, 6 ml bolus dose and 30 min lockout time will be performed till 48 h postoperative period.
  Interventions: Other: ESP block (Group A)
- Group TEA = Thoracic epidural analgesia group (Active Comparator): TEA will be performed in the preoperative block room.A continuous infusion of 0.125% bupivacaine at the rate of 4 ml/h infusion dose, 6 ml bolus dose and 30 min lockout time will be performed till 48 h postoperative period.
  Interventions: Other: TEA group (Group B)

INTERVENTIONS:
Other: ESP block (Group A) — US probe will be placed longitudinally 2-3 cm lateral to the T5 transvers process. From superior to inferior, three muscles will be visualized on the hyperechoic transverse process; trapezius (upper), rhomboideus major (middle), erector spinae (lower). The block needle will be inserted cranio caudal direction and then for correction of the needle 5 ml saline will be injected deep into the erector spina muscle fascia. Following confirmation of the correct position 20G catheter will be inserted 5 cm in caudal direction. 20 ml %0.25 bupivacaine will be administered for block.
  Arms: Group ESPB = Erector spinae plane block group
Other: TEA group (Group B) — Local infiltration with 2% of lidocaine under the skin, in T4/T5 intervertebral space will be administered. An 18 G Tuohy needle will be inserted at T4/T5 intervertebral space to identify epidural space using the loss of resistance technique. 20G catheter will be inserted 3-4 cm in caudal direction in the epidural space. Bolus dose of 0.125% bupivacaine 10 ml will be administered through the catheter after the negative aspiration for blood or cerebrospinal fluid
  Arms: Group TEA = Thoracic epidural analgesia group

SUMMARY:
Video assisted thoracic surgery (VATS) has recently been evaluated as the standard surgical procedure for lung surgery. Although VATS is less painful than thoracotomy, patients may feel severe pain during the first hours at postoperative period. Analgesia management is very important for these patients in postoperative period since insufficient analgesia can cause pulmonary complications such as atelectasis, pneumonia and increased oxygen consumption. The ultrasound (US) guided erector spina plane (ESP) block is a novel interfacial plan block defined by Forero et al. at 2016. ESP block provides thoracic analgesia at T5 level and abdominal analgesia at T7-9 level. Visualization of sonoanatomy with US is easy, and the spread of local anesthesic agents can be easily seen under the erector spinae muscle (12). Thus, analgesia occurs in several dermatomes with cephalad-caudad way. In the literature, there is not still any randomized study evaluating ESP block efficiency for postoperative analgesia management after VATS. The aim of this study is to compare US-guided continuous ESP block and TEA for postoperative analgesia management after VATS.

DETAILED DESCRIPTION:
Video assisted thoracic surgery (VATS) has recently been evaluated as the standard surgical procedure for lung surgery. The advantages of VATS procedures compared with open thoracotomy are rapid recovery, short hospital stay and low complication risk. Although VATS is less painful than thoracotomy, patients may feel severe pain during the first hours at postoperative period. Thoracic epidural analgesia (TEA) which is the gold standard analgesic technique after thoracotomy, is generally used for analgesia management after VATS. However, since the surgical technique and trauma between open surgery and VATS are different, the question of what should be the gold standard for analgesia management after VATS is a topic of discussion. Especially due to the difficult administration and adverse effect profile of TEA, the opinion of minimally invasive surgical procedures, requiring less invasive analgesic techniques is supported. Analgesia management is very important for these patients in postoperative period since insufficient analgesia can cause pulmonary complications such as atelectasis, pneumonia and increased oxygen consumption.

The ultrasound (US) guided erector spina plane (ESP) block is a novel interfacial plan block defined by Forero et al. at 2016. ESP block provides thoracic analgesia at T5 level and abdominal analgesia at T7-9 level. The ESP block contains a local anesthetic injection into the deep fascia of erector spinae. This area is away from the pleural and neurological structures and thus minimizes the risk of complications due to injury. Visualization of sonoanatomy with US is easy, and the spread of local anesthesic agents can be easily seen under the erector spinae muscle. Thus, analgesia occurs in several dermatomes with cephalad-caudad way. Cadaveric studies have shown that the injection spreads to the ventral and dorsal roots of the spinal nerves and creates sensory blockade in both posterior and anterolateral thorax. In the literature, it has been reported that ESP block provides effective analgesia after open heart surgery, breast surgery and ventral hernia repair in randomized controlled studies about ESP block efficiency for postoperative analgesia management. In some case series and case reports it has been reported that ESP block provides effective analgesia after thoracotomy and VATS. Furthermore, it has been reported that it provides effective analgesia in chronic and persistant pain syndromes of thorax.

The aim of this study is to compare US-guided continuous ESP block and TEA for postoperative analgesia management after VATS. The primary aim is to compare perioperative and postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), adverse effects related with opioids (allergic reaction, nausea, vomiting), complications due to blocks (pneumothorax, hematoma), and the time period and number of attempt for blocks.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for lVATS under general anesthesia

Exclusion Criteria:

* Bleeding diathesis
* Receiving anticoagulant treatment
* Known local anesthetics and opioid allergy
* Infection of the skin at the site of the needle puncture
* Pregnancy or lactation
* Patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores | Postoperative 24 hours
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores at rest and during cough will be recorded at postoperative 0, 2, 4, 8, 16,and 24 hours.

SECONDARY OUTCOMES:
Rescue analgesia need | Postoperative 0, 2, 4, 8, 16, and 24 hours.
  Postoperative rescue analgesia need will be evaluated at postoperative 0, 2, 4, 8, 16, and 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Bahadir Ciftci, Asist.Prof, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Continuous Erector Spinae Plane Block for Rescue Analgesia in Thoracotomy After Epidural Failure: A Case Report. A A Case Rep. 2017 May 15;8(10):254-256. doi: 10.1213/XAA.0000000000000478. PMID 28252539
- [Background] Nagaraja PS, Ragavendran S, Singh NG, Asai O, Bhavya G, Manjunath N, Rajesh K. Comparison of continuous thoracic epidural analgesia with bilateral erector spinae plane block for perioperative pain management in cardiac surgery. Ann Card Anaesth. 2018 Jul-Sep;21(3):323-327. doi: 10.4103/aca.ACA_16_18. PMID 30052229
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005